CLINICAL TRIAL: NCT00995839
Title: Vasopressin Receptor Agonists in Septic Shock: Effects on Microcirculation
Brief Title: Terlipressin in Septic Shock: Effects on Microcirculation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Andrea Morelli, University of Rome "La Sapienza"
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1065
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2009-10

CONDITIONS: Septic Shock; Sepsis
Keywords: terlipressin; vasopressin; sepsis; septic shock; norepinephrine
MeSH Terms: conditions — Shock, Septic; Sepsis; Diabetes Insipidus | interventions — Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- continuous terlipressin (Experimental)
  Interventions: Drug: continuous infusion of terlipressin
- vasopressin (Experimental)
  Interventions: Drug: Arginine vasopressin
- terlipressin bolus dose (Experimental)
  Interventions: Drug: terlipressin bolus administration

INTERVENTIONS:
Drug: continuous infusion of terlipressin — Intravenous continuous infusion of terlipressin 1 µg•kg-1•h-1 for 6 hrs
  Arms: continuous terlipressin
Drug: Arginine vasopressin — Intravenous continuous infusion of arginine vasopressin 0.04 UI•min-1 for 6 hrs
  Arms: vasopressin
Drug: terlipressin bolus administration — intravenous terlipressin bolus administration at the dose of 0.5 mg
  Arms: terlipressin bolus dose

SUMMARY:
The present study was conducted as a prospective, randomized study to investigate the effects of vasopressin receptor agonists terlipressin and vasopressin on systemic hemodynamics and microcirculation in patients with catecholamine-dependent septic shock.

DETAILED DESCRIPTION:
60 septic shock patients requiring norepinephrine to maintain mean arterial pressure between 65 and 75 mmHg despite adequate volume resuscitation will be enrolled in the study. After an initial hemodynamic resuscitation aimed at achieve a mean arterial pressure between 65 and 75 mmHg and normovolemia, patients will be randomly allocated to be treated with either a) intravenous administration of terlipressin 1 µg∙kg-1∙h-1 for 6 hrs, b) intravenous administration of arginine vasopressin 0.04 UI∙min-1 for 6 hrs, c) intravenous administration of terlipressin bolus dose of 0.5 mg (each n = 20). In all groups open label norepinephrine will be additionally administered to maintain a mean arterial pressure (MAP) between 65 and 75 mmHg, if necessary. Data from right heart catheterization and sublingual microvascular network will be obtained just before randomization (baseline) and then after 6 hours in the vasopressin, terlipressin infusion and terlipressin bolus groups.

The sublingual microvascular network will be studied using the sidestream dark field (SDF)imaging. The device will be applied on the lateral side of the tongue, in an area approximately 2-4 cm from the tip of the tongue. Sequences of 10 secs from eight adjacent areas will be recorded on disk using a personal computer. These sequences will be later analyzed by an investigator blinded to the patient's diagnosis and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of septic shock
* Vasopressor support to maintain mean arterial pressure (MAP) between 65 and 75 mmHg despite adequate volume resuscitation (pulmonary artery occlusion pressure = 13-18 mmHg and central venous pressure = 8-12 mmHg)

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* Present or suspected acute mesenteric ischemia
* Vasospastic diathesis (e.g. Raynaud's syndrome or related diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Systemic hemodynamic and Microcirculatory flow index of small and medium vessels (MFI) | over a period of 6 hrs from the time of randomization
Oxygen transport variables | over a period of 6 from the time of randomization

SECONDARY OUTCOMES:
Acid-base homeostasis | over a period of 6 hrs from the time of randomization
Functional capillary density (mm/mm2) (FCD) | over a period of 6 hrs from the time of randomization
De Backer score | over a period of 6 hrs from the time of randomization
Perfused Vessel Density (PVD) (mm/mm2) | over a period of 6 hrs from the time of randomization
Proportion of Perfused vessels (%) (PPV) | over a period of 6 hrs from the time of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Principal Investigator — University of Rome "La Sapienza", Department of Anesthesiology and Intensive Care
Locations (1):
- Departement of Anesthesiology and Intensive Care, Rome, I, Italy

REFERENCES:
- [Derived] Morelli A, Donati A, Ertmer C, Rehberg S, Kampmeier T, Orecchioni A, Di Russo A, D'Egidio A, Landoni G, Lombrano MR, Botticelli L, Valentini A, Zangrillo A, Pietropaoli P, Westphal M. Effects of vasopressinergic receptor agonists on sublingual microcirculation in norepinephrine-dependent septic shock. Crit Care. 2011;15(5):R217. doi: 10.1186/cc10453. Epub 2011 Sep 19. PMID 21929764